CLINICAL TRIAL: NCT06316739
Title: Ending HIV and Taming Hepatitis C Virus and Overdose Among Puerto Rican People Who Inject Drugs in New York City: The Ganchero Intervention
Brief Title: The Ganchero Intervention for Migrant People Who Inject Drugs From Puerto Rico in New York City
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: North Jersey AIDS Alliance dba North Jersey Community Research Initiative (NJCRI) (Other)
Collaborators: City University of New York, School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R34DA057166 (NIH)
Record Dates: First submitted 2024-02-27; First posted 2024-03-18 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections; HCV; Overdose
Keywords: people who inject drugs (PWID); Puerto Ricans; peer intervention; HIV prevention; injection drug use; naloxone
MeSH Terms: conditions — HIV Infections; Drug Overdose

STUDY DESIGN:
Intervention Model Description: Non-randomized wait-list controlled trial. The intervention will be implemented in 2 neighborhoods (in the Bronx, New York City) sequentially. Outcomes among participants in the immediate intervention neighborhood will be compared to outcomes among participants in the delayed intervention neighborhood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention neighborhood (Experimental): According to the trial's wait-list controlled design, the Ganchero intervention will be implemented sequentially in two geographically and socially distinct Bronx neighborhoods with large migrant Puerto Rican populations. In Cycle I, the intervention will be implemented with Gancheros and their clients in neighborhood A, while participants in neighborhood B receive standard access to harm reduction through a local Syringe Services Program (SSP).
  Interventions: Behavioral: Ganchero intervention
- Delayed intervention neighborhood (Experimental): In Cycle II, the Ganchero intervention will be implemented with Gancheros and their clients in neighborhood B, while participants in neighborhood A receive standard access to harm reduction through a local Syringe Services Program (SSP).
  Interventions: Behavioral: Ganchero intervention

INTERVENTIONS:
Behavioral: Ganchero intervention — The Ganchero intervention is an HIV, hepatitis C virus (HCV) and overdose prevention intervention for migrant people who inject drugs (PWID) from Puerto Rico who are living in New York City. The intervention has two core components, both centered around the key migrant PWID role of the "Ganchero," an individual who provides expert injection services in exchange for money or drugs. First, a sample of Gancheros will be trained in foundational HIV, HCV and overdose risk-reduction knowledge and outreach strategies (over 6 2-hour, in-person, small group sessions facilitated by an Interventionist). Second, during a 4-month outreach period, trained Gancheros will disseminate risk-reduction messages learned in the training, and associated resources (e.g., sterile syringes and other injection equipment, naloxone), to migrant PWID in their neighborhood as they deliver their regular Ganchero services.

SUMMARY:
The goal of this pilot clinical trial is to learn if an intervention that trains Gancheros (people who provide injection services in exchange for drugs or money) to conduct risk-reduction outreach could help lower risk for human immunodeficiency virus (HIV), hepatitis C virus (HCV) and overdose among migrant Puerto Rican people who inject drugs (PWID) in New York City. The main questions it aims to answer are:

* Can the Ganchero intervention be carried out successfully and will Gancheros and their clients like it?
* Could the Ganchero intervention help Puerto Rican PWID who are clients of Gancheros use sterile syringes and carry naloxone (a medication to reverse opioid overdoses) more often?

Gancheros who participate in the trial will be asked to attend a 6-session training on HIV, HCV, and overdose prevention and then to share key prevention messages and supplies (e.g., naloxone, sterile syringes and other injection equipment) with their clients during 4 months of outreach. The intervention will be carried out with Gancheros and their clients in two Bronx neighborhoods, one after the other, so the investigators can see if clients in the neighborhood that received the intervention first have better outcomes than clients in the neighborhood that did not yet receive the intervention.

DETAILED DESCRIPTION:
The threat of human immunodeficiency virus (HIV) among people who inject drugs (PWID) in New York City (NYC) is not over. Multiple HIV outbreaks among PWID in rural and urban areas of the United States (US) have occurred recently, from 2015 in rural Indiana to 2018 in northeastern Massachusetts. PWID who are racial/ethnic minorities continue to be disproportionately infected with HIV. Among these, Puerto Rican (PR) PWID who started injecting drugs in Puerto Rico and continue to inject drugs in NYC remain highly vulnerable not only to HIV, but also to hepatitis C virus (HCV) and fatal opioid overdose. Analyses of two different cycles of the National HIV Behavioral Surveillance (NHBS) study conducted by the Centers for Disease Control and Prevention (CDC) in NYC found PR PWID, especially those who migrated from Puerto Rico, to be the most HIV-vulnerable ethnic group. In 2017, the US overdose mortality rate for US-born and Puerto Rico-born PR PWID exceeded the rate for Non-Hispanic Whites, and the same holds true in NYC. Recent research showed that PR PWID (both US- and Puerto Rico-born) have significantly higher prevalence of HCV than non-PR-PWID, and that Puerto Rico-born migrant PWID have the highest HCV prevalence (86%) of all three groups. Consequently, helping Puerto Rico-born PWID avoid HIV will help prevent HIV outbreaks in NYC. Lowering their HCV and overdose risk will help reduce overall HCV prevalence (67%) and overdose mortality rates (21.2 per 100,000) in NYC's PWID. Meeting these goals is urgent, as PWID migration from Puerto Rico to NYC is ongoing, as evidenced by their sizeable (≥25%) presence in NHBS studies in the past 15 years.

Risk behaviors of migrant PR PWID in the US are well documented. Compared to non-migrant PWID, migrants regularly engage in syringe- and cooker-sharing. In NYC, PR migrants mostly reside in the Bronx, the county with the largest numbers of PWID, overdose deaths, and new cases of HIV, and very high HCV prevalence in PWID. In a recent National Institute for Drug Abuse (NIDA)-funded ethnographic study (R03DA041892), the Principal Investigators identified normative practices learned while injecting drugs in Puerto Rico as critical influences on migrants' risks in NYC. These practices include: pervasive syringe-sharing after "cleaning" syringes by "air-blowing and water-rinsing"; regular sharing and trading of heavily used cookers which are highly valued for their concentrated drug residue; and low rates of naloxone carriage despite frequent overdoses.

Grounded in a multi-level ecosocial framework, the proposed intervention will directly target these practices by leveraging a key migrant PWID-role in NYC, the Ganchero: an "injection doctor" who exchanges injection expertise for drugs or money. Because migrant PWID regularly require expert injection services due to collapsed veins, Gancheros are central network members well-positioned to promote positive health change. This is aligned with social network diffusion theory, which underlies effective HIV prevention interventions that harness peer influence by relying on PWID to disseminate risk-reduction messages in their networks. PR migrant PWID are highly networked, and a peer-driven intervention relying on their network ties promises to yield sustainable health behavior change. The investigators will develop and conduct an initial evaluation of a Ganchero risk-reduction intervention for Puerto Rico-born PWID that is effective, culturally appropriate, credible, and sustainable.

First, a multi-method, iterative process that will incorporate input from Gancheros and their migrant clients will be used to develop the intervention: a training curriculum and outreach protocol for Gancheros. Building on specific intervention recommendations developed in consultation with a multiple-stakeholder Intervention Advisory Board and endorsed by focus groups of migrant PWID in the investigators' prior study, the intervention will empower Gancheros to promote and model consistent sterile syringe use and naloxone carriage with their clients and in their PWID networks. Targeting two Bronx neighborhoods with high proportions of PR migrants and non-overlapping PWID networks, the investigators will then conduct a pilot clinical trial to evaluate the feasibility, acceptability, and preliminary effectiveness of this innovative intervention.

Aim 1. Engage Gancheros (total n=4) and clients (total n=20) from both target neighborhoods in a series of semi-structured interviews and focus groups to develop a risk-reduction intervention comprised of a training curriculum and outreach protocol for Gancheros to implement with their regular clients in real-world settings.

Aim 2. Conduct a pilot clinical trial using a wait-list control design with 10 Gancheros and 60 clients across the two target neighborhoods to evaluate the intervention's feasibility (assessed via Ganchero and client participation rates), acceptability (assessed by Ganchero and client Visual Analog Scale [VAS] ratings and qualitative feedback) and preliminary effectiveness in increasing clients' rates of sterile syringe use (primary effectiveness outcome) and naloxone carriage (secondary effectiveness outcome).

Structured assessments to measure these outcomes will be supplemented with data from Gancheros' Weekly Outreach Reports and systematic ethnographic observations of Gancheros deploying intervention strategies in the field to assess fidelity of implementation, barriers encountered, and any pragmatic adaptations made in response to barriers, to inform future refinement of the intervention and its implementation strategy.

Impact: A Ganchero-led intervention may help prevent HIV outbreaks among PWID in NYC and mitigate the HCV and overdose syndemic among the highly vulnerable Puerto Rico-born PWID in NYC. Results will inform a larger hybrid effectiveness-implementation trial to evaluate a refined intervention for migrant PR PWID in NYC and other urban areas in the US with significant numbers of at-risk migrants.

ELIGIBILITY:
Two distinct groups of participants with different eligibility criteria will be enrolled: (1) Gancheros (n=10, 5/neighborhood); and (2) Gancheros' clients (n=60, 30/neighborhood).

1. Ganchero participants:

   * Inclusion Criteria:

     * A migrant person who injects drugs (PWID) from Puerto Rico living in one of 2 pre-selected neighborhoods in the Bronx, New York City (NYC)
     * Past experience providing Ganchero services in Puerto Rico
     * Currently provides Ganchero services to ≥10 clients/day
     * Speaks Spanish or English
   * Exclusion Criteria:

     * Planned travel away from NYC for 2 weeks or longer over the next 24 months
     * Inability to comprehend trial information or provide informed consent (e.g., due to intoxication)
2. Client participants:

   * Inclusion Criteria:

     * A migrant PWID from Puerto Rico living in one of 2 pre-selected neighborhoods in the Bronx, NYC
     * Referred to the study by a participating Ganchero
     * Used the services of their nominating Ganchero at least once/week for the past 90 days
     * Speaks Spanish or English
   * Exclusion Criteria:

     * Inability to comprehend trial information or provide informed consent (e.g., due to intoxication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
sterile syringe use | past 30 days; assessed at the end of Cycle I (each Cycle is a total of 7 months long)
  number of sterile syringes per day each client reports using, with an offset term for the number of injections per day

SECONDARY OUTCOMES:
naloxone carriage | past 30 days; assessed at the end of Cycle I (each Cycle is a total of 7 months long)
  number of days per week each client reports carrying naloxone

OTHER OUTCOMES:
Feasibility of intervention - Ganchero Engagement | 7 months
  Gancheros' attendance at 6 training sessions and 16 weekly meetings with Interventionist during outreach period
Feasibility of intervention - Client Engagement | 4 months
  Mean number of clients engaged/day by all participating Gancheros during 4-month outreach period
Acceptability of the intervention's training component to Gancheros | 3 weeks, assessed at the end of the Ganchero training which will consist of 6 sessions scheduled over 3 weeks
  Average score across 10 0-100mm visual analog scale (VAS) items (anchored by 0-Not at all and 100-A great deal) regarding specific attributes of the Gancheros' HIV, HCV and overdose training, such as: its likeability; the effectiveness and relatability of the Interventionist/trainer; the usefulness and comprehensibility of the didactic content, including the safer drug use/injection practices presented; its relevance to the drug use and injection practices of migrant PWID; and the usefulness of the interactive activities and exercises.
Acceptability of the intervention's outreach component to Gancheros | 4 months
  Average score across 10 0-100mm visual analog scale (VAS) items (anchored by 0-Not at all and 100-A great deal) regarding specific aspects of the outreach protocol for Gancheros, such as: the extent to which the training prepared them to conduct risk-reduction outreach in their community; the usefulness and sufficiency of the harm reduction supplies and other resources provided; and the usefulness and sufficiency of the support provided to help Gancheros overcome barriers encountered in the field.
Acceptability of intervention to Clients | 4 months
  Average score across 10 0-100mm visual analog scale (VAS) items (anchored by 0-Not at all and 100-A great deal) regarding specific attributes of the intervention such as its likeability, usefulness in promoting safer drug use/injection practices, and relevance to the lives of migrant PWID; the ease of implementing its risk-reduction strategies; the credibility of Gancheros as harm reduction peer leaders; the extent to which it fostered a sense of community empowerment; and the sustainability of behavioral changes spurred by the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- CUNY Graduate School of Public Health & Health Policy, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided